CLINICAL TRIAL: NCT00712517
Title: Do Patients Anesthetized With Propofol Have Less Pain Than Those Anesthetized With Volatile?
Brief Title: Propofol Versus Volatile Anesthesia in Post Operative Pain Management
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Enrolling of participants has halted and the results are being gathered
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 42908
Record Dates: First submitted 2008-07-07; First posted 2008-07-10 (Estimated); Last update posted 2016-07-20 (Estimated); Status verified 2016-07

CONDITIONS: Varicose Vein; Postoperative Pain
Keywords: postoperative pain; Piritramid; propofol; sevoflurane; varicose vein; Anesthesia
MeSH Terms: conditions — Varicose Veins; Pain, Postoperative | interventions — Propofol; Sevoflurane

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Patients will receive propofol anesthesia during varicose vein stripping surgery.
  Interventions: Drug: propofol
- 2 (Active Comparator): Patients will receive sevoflurane anesthesia during varicose vein stripping surgery.
  Interventions: Drug: sevoflurane

INTERVENTIONS:
Drug: propofol — propofol anesthesia 3-5mg/kg
  Other Names: Diprivan
  Arms: 1
Drug: sevoflurane — sevoflurane anesthesia
  Arms: 2

SUMMARY:
The study will test the hypothesis that patients anesthetized with propofol suffer less postoperative pain than those anesthetized with sevoflurane.

DETAILED DESCRIPTION:
Patients undergoing s stripping operation for varicose veins will be randomized to one of two groups. Group 1 patients will receive propofol anesthesia. Group 2 patients will receive sevoflurane anesthesia. Intraoperative measurements including mean-arterial pressure, heart rate, propofol infusion rate, remifentanil infusion rate, and end-tidal sevoflurane concentration will be taken at 15 minute intervals. Patients in both groups will receive Piritramid as necessary to control pain either intravenously or through patient controlled pump. VAS pain score, mean-arterial pressure, heart rate, nausea will be evaluated at 30 minute intervals during the first four postoperative hours. Piritramid dosage and vomiting will be recorded through the first postoperative morning. Patients will rate pain based on the VAS score for the period between leaving the recovery room and the first postoperative morning

ELIGIBILITY:
Inclusion Criteria:

* Participants will undergo a stripping operation for varicose veins
* Surgery will be performed by one physician only
* Written informed consent

Exclusion Criteria:

* Any contraindications to the proposed interventions
* Procedures done under regional anesthesia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2010-09; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
The primary outcome is morphine-equivalent use from the end of surgery until the first post-operative morning. | first post operative morning

SECONDARY OUTCOMES:
To determine the average pain score for each group during the first four hours of recovery after surgery. | 30 minute intervals for first 4 hours post operatively

CONTACTS AND LOCATIONS:
Overall Officials: Olga Plattner, MD, Principal Investigator — Medical University of Vienna
Locations (1):
- Olga Plattner , MD, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Windpassinger M, Plattner O, Gemeiner J, Bohler K, Luntzer R, Klimscha W, Yang D, Mascha EJ, Sessler DI. Opioid use after propofol or sevoflurane anesthesia: a randomized trial. Can J Anaesth. 2016 Nov;63(11):1258-65. doi: 10.1007/s12630-016-0728-5. Epub 2016 Sep 14. PMID 27638296